CLINICAL TRIAL: NCT01466075
Title: Clinical Study of the Apollo Evolution BGMS With Tatsu Blood Glucose Test Strips
Brief Title: Study of an Investigational Glucose Meter System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R&D-2011-2012-0.03
Record Dates: First submitted 2011-10-28; First posted 2011-11-07 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the Monitoring System (Experimental): Untrained subjects with diabetes use the Apollo Evolution Investigational BG Monitoring System.
  Interventions: Device: Apollo Evolution Investigational BG Monitoring System

INTERVENTIONS:
Device: Apollo Evolution Investigational BG Monitoring System — Untrained subjects with diabetes perform self Blood Glucose (BG) tests with capillary fingerstick blood and Alternative Site Testing (AST) of the palm using the Apollo Evolution meter and an investigational sensor. Study staff test subject venous blood and all BG results are compared to a reference laboratory glucose method. Untrained subjects complete basic tasks using the User Guide and provide feedback.

SUMMARY:
The purpose of this study is to demonstrate that untrained subjects who have diabetes or pre-diabetes can operate the investigational Blood Glucose Monitoring System (BGMS) and obtain valid glucose results.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of diabetes or pre-diabetes.
* Be 18 years of age or older
* Be able to speak, read and understand English and understand the Informed Consent document.
* Be willing to complete study procedures

Exclusion Criteria:

* Pregnancy
* Infections or skin disorders at the site of the venipuncture (at the discretion of the phlebotomist).
* Hemophilia, bleeding disorder, or clotting problems. Persons taking aspirin (81 mg or 325 mg) daily or Plavix® are not reason for exclusion.
* Physical (dexterity), visual, or neurological impairments that would make the person unable to perform testing with the BGM (at the discretion of the site professional staff).
* A condition, in the opinion of the Investigator, would put the subject at risk or influence the conduct of the study or interpretation of the results. The reason for exclusion will be documented by the professional staff.
* Previously participated in a blood glucose monitoring study using a similar device or use a similar device for personal use when monitoring blood glucose.
* Working for a competitive medical device company or having an immediate family member or someone who is not a family member but is living within the household of someone who works for such a company
* Working for a medical laboratory, hospital or other clinical setting that involves training on and clinical use of blood glucose monitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Simmons, MD, Principal Investigator — Ascensia Diabetes Care
Locations (1):
- Bayer HealthCare LLC, Diabetes Care, Mishawaka, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intended Users of the Monitoring System: Untrained subjects with diabetes use the Apollo Evolution Investigational Blood Glucose Monitoring System.
  Apollo Evolution Investigational BG Monitoring System : Untrained subjects with diabetes perform self Blood Glucose (BG) tests with capillary fingerstick blood and AST of the palm using the Apollo Evolution meter and an investigational sensor. Study staff test subject venous blood. All BG results are compared to a reference laboratory glucose method. Untrained subjects complete basic tasks using the User Guide and provide feedback.
Period: Overall Study
Arm/Group | Intended Users of the Monitoring System
Started | 207
Completed | 207
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 207
Age, Continuous [Mean (Full Range); unit: years] | 55.7 [18 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117
  Male | 90
Region of Enrollment [Number; unit: participants]
  United States | 207

OUTCOME MEASURES:

1. Primary Outcome: Percent of Self-Test Fingerstick Blood Glucose Results Within +/- 15mg/dL (<75mg/dL) or Within +/- 20% (>=75mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-test fingerstick blood using the Apollo Evolution Investigational Blood Glucose Monitoring System (BGMS). BGMS results are compared with capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results are used to calculate the number of BGMS results within +/- 15mg/dL (<75mg/dL YSI capillary plasma) or +/- 20% (>=75mg/dL YSI capillary plasma). Site staff tested in parallel after subjects.
Time Frame: 1 hour
Population: Blood data for three subjects were not evaluable because the difference between the replicates of the reference YSI analyzer measurements exceeded the protocol defined criteria. Remaining 204 subjects each tested one of three test strip lots on the system. 204 (207-3) test results were available.
Measure: Number; unit: percentage of Blood Glucose Test Results
Units Other Than Participants: Blood Glucose Test Results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 204
Number analyzed (Blood Glucose Test Results) | 204
percentage of Blood Glucose Test Results | 99.51

2. Secondary Outcome: Percent of Glucose Results From Alternative Site Testing (AST) of the Palm Within +/- 15mg/dL (<75mg/dL) or Within +/- 20% (>=75mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-test Alternative Site (AST) Palm blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS AST results are compared with capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI capillary plasma BG results are used to calculate the number of AST BGMS results within +/- 15mg/dL (<75mg/dL YSI capillary plasma) or +/- 20% (>=75mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: Blood data for three subjects were not evaluable because the difference between the replicates of the reference YSI analyzer measurements exceeded the protocol defined criteria. The remaining 204 subjects each tested one of three test strip lots on the system. 204 (207-3) test results were available.
Measure: Number; unit: percentage of Blood Glucose Test Results
Units Other Than Participants: Blood Glucose Test Results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 204
Number analyzed (Blood Glucose Test Results) | 204
percentage of Blood Glucose Test Results | 99.51

3. Secondary Outcome: Percent of Venous Blood Glucose Results Within +/- 15mg/dL (<75mg/dL) or Within +/- 20% (>=75mg/dL) of Laboratory Glucose Method
Description: Study staff tested subject venous blood using an investigational Blood Glucose Monitoring System (BGMS). Venous BGMS results are compared with venous plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI venous plasma results are used to calculate the number of BGMS results within +/- 15mg/dL (<75mg/dL YSI venous plasma) or +/- 20% (>=75mg/dL YSI venous plasma).
Time Frame: 1 hour
Population: 609 venous BG results(203 subjects x 3 test strip lots) were available. Three subjects did not have successful venipunctures so no blood obtained. BGMS testing was not performed with one subject's blood sample. Study staff tested each subject venous blood sample using 3 test strip lots.
Measure: Number; unit: percentage of Blood Glucose Test Results
Units Other Than Participants: Venous BG Test Results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 203
Number analyzed (Venous BG Test Results) | 609
percentage of Blood Glucose Test Results | 100.0

4. Secondary Outcome: Number of Subjects Able to Perform Given Tasks Using Product Labeling for Instruction
Description: After reading the instructions for use, and without assistance from the study staff, subjects use the BGMS to perform basic tasks considered to be essential for the operation of the system.
Time Frame: 1 hour
Population: Blood data for three subjects were not considered evaluable because the difference between the replicates of the reference YSI analyzer measurements exceeded the protocol defined criteria. Remaining 204 subjects each tested one of three test strip lots on the system. 204 (207-3) test results were available.
Measure: Number; unit: participants
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 204
participants
  Successfully performed fingerstick BG test | 203
  Successfully performed palm AST BG test | 203

ADVERSE EVENTS:
Arm/Group | Intended Users of the Monitoring System
Serious Adverse Events (participants affected / at risk) | 0/207
Other Adverse Events (participants affected / at risk) | 1/207
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intended Users of the Monitoring System (N=207)
hypoglycemia (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No